CLINICAL TRIAL: NCT00429728
Title: An Open-Label, Parallel Group, Single Session Study Comparing the Pharmacokinetics of a Single Oral Dose of GW876008 Administered to Healthy Volunteer Smokers and Healthy Volunteer Non-Smokers.
Brief Title: A Study To Investigate The Metabolism Of GW876008 In Smokers Compared To Non-Smokers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRH103004
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics,; tolerability,; healthy,; subjects,; smokers,; non-smokers
MeSH Terms: interventions — GW 876008

INTERVENTIONS:
Drug: GW876008

SUMMARY:
This study will investigate the effect of smoking on the metabolism of a single oral dose of GW876008.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females.
* Normal ECG.
* Non-smokers (abstinence from smoking for at least 6 months before the start of the study) or smokers who smoke between 10 and 30 cigarettes, inclusive, per day, for at least 2 months prior to screening.
* Subjects must agree to abstain from alcohol for 24 hours prior to the start of dosing until collection of the final pharmacokinetic sample.

Exclusion Criteria:

* Any serious medical disorder or condition.
* Any clinically significant laboratory abnormality.
* History of psychiatric illness.
* Any history of suicidal attempts or behavior.
* Active peptic ulcer disease.
* Positive faecal occult blood.
* Current or recent (within one year) gastrointestinal disease; a history of malabsorption, oesophageal reflux, irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn; or any surgical intervention (e.g., cholecystectomy) which would be expected to influence the absorption of drugs.
* Female subjects who are currently or who are planning to become pregnant or who are lactating (from screening through at least 8 weeks after receiving study drug).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-11

PRIMARY OUTCOMES:
Blood levels of GW876008 collected on Day 1 at pre-dose and over 72 hours post-dose. | on Day 1 at pre-dose and over 72 hours post-dose.

SECONDARY OUTCOMES:
12-lead ECG on day 1, 24 hours post dose, & follow up | on day 1, 24 hours post dose, & follow up
vital signs at screening & day 1 through 72 hours post dose | at screening & day 1 through 72 hours post dose
adverse events day 1 through 72 hours post dose | day 1 through 72 hours post dose
clinical laboratory data day 1 through 24 hours post dose | day 1 through 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MBChB, MFPM, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Willingboro, New Jersey, United States